CLINICAL TRIAL: NCT07220863
Title: Evaluation of the Safety and Efficacy of a Wearable Device Based on Thermometry and Impedance Technology for Breast Mapping and Detecting Suspicious Breast Lesions Using Feminai 1.0
Brief Title: Breast Mapping and Detection of Suspicious Breast Lesions Using Feminai
Status: Recruiting | Type: Observational
Sponsor: Feminai (Industry)
Responsible Party: Sponsor
Other Study IDs: 03-FLTD
Record Dates: First submitted 2025-10-21; First posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer Awareness
Keywords: Breast lesions; Breast mapping; Home breast examination; Wearable patch; Thermometry; Bioimpedance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- breast cancer screening: Women between the ages 25-75 undergoing breast cancer screening

SUMMARY:
Prospective observational study evaluating the safety and accuracy of Feminai 1.0, an at-home adhesive patch that measures skin temperature and electrical impedance to map each breast. Up to 300 women (ages 25-75) undergoing screening will have one study visit; Feminai results will be compared with mammography and, when available, biopsy to assess sensitivity and negative predictive value. Feminai is investigational, intended to support clinical decision-making, and does not replace standard diagnostic tests.

DETAILED DESCRIPTION:
This study will evaluate Feminai 1.0, a home breast examination kit that uses skin-surface temperature and electrical impedance measurements to create a "map" of each breast. The goal is to learn whether Feminai can help identify the presence or absence of suspicious soft-tissue lesions that may need further medical evaluation. The device is intended to support clinical decision-making and is not a stand-alone diagnostic test.

Who can join:

Women ages 25-75 who are undergoing breast cancer screening. Two groups will be enrolled:

* About 150 women whose most recent screening mammogram was read as low concern (similar to BI-RADS 1-2).
* About 150 women who are scheduled for a biopsy after a mammogram that showed higher concern (similar to BI-RADS 4-5).

Key exclusions include current treatment for breast cancer, pregnancy or breastfeeding, metal implants, recent breast surgery (within 1 year), breast implants/injections, cup size larger than US size E, and any condition that would make participation unsafe or impractical.

What participation involves:

This is a prospective, observational study with one visit. After informed consent and eligibility confirmation, trained staff will apply the Feminai patch in a private room to collect measurements from each breast. Participants will complete a short questionnaire about their experience. Routine clinical care (such as mammography and, if planned, biopsy) will occur as usual; there is no randomization and no change to standard care. To avoid anxiety or influencing medical decisions, Feminai results will not be shared with participants or their physicians.

Risks and discomforts:

Expected risks are minor and temporary, similar to other adhesive skin patches: mild skin redness or irritation, itching, slight discomfort when the patch is removed, brief indentation marks, or mild dryness/sensitivity, especially with repeated applications. Serious device-related risks are not expected but will be monitored. Any device malfunctions will be recorded.

ELIGIBILITY:
Inclusion Criteria:

General:

1. Females aged 25-75 years.
2. Able to comply with study procedures and follow-up requirements.
3. Willing and able to provide informed consent.

Additional for Group 1 (up to N=150):

1. Presenting for routine mammography/tomosynthesis breast cancer screening according to national/regional guidelines.
2. Most recent mammography result - BIRADS 1 or 2

Additional for Group 2 (up to N=150):

1. Presenting for biopsy following BIRADS 4-5 mammogram

Exclusion Criteria:

1. History of current treatment for breast cancer.
2. Pregnancy or lactation.
3. Presence of any implanted metal.
4. Any condition that, in the opinion of the investigator, may interfere with the participant's ability to comply with study requirements or may pose a risk to the participant.
5. Has breast enhancements (e.g. implants or injections)
6. Subjects who have undergone surgery (e.g. lumpectomy or mastectomy) in the last year at the time of study enrollment
7. No subject will be allowed to enroll in this trial more than once.
8. Cup size larger than E in US-based sizing charts.

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Women between the ages 25-75 undergoing breast cancer screening
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-05 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2026-09-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and NPV | From enrollment to the time the the ground truth is available followed for up to 6 months
Sensitivity and NPV | From enrollment to the time that the mammography and biopsy results (if applicable) are available followed for up to 6 months.
  The co-primary endpoints will be defined on a per patient basis as sensitivity and NPV. The endpoints will be based on the binary outcomes produced for each breast side (right and left).
  For side-level analysis, the definitions of True Positive (TP), False Positive (FP), True Negative (TN), and False Negative (FN) are as follows:
  TP side: Side is Ground Truth (GT) positive and Flagged by device FP side: Side is GT negative and Flagged by device FN side: Side is GT positive and Not Flagged by device TN side: Side is GT negative and Not Flagged by device
  For subject-level analysis, the definitions of TP, FP, TN, and FN are based on side-level classification, as follows:
  TP subject: A subject has only one GT positive side and this side is Flagged by the device. Or, a subject has 2 GT positive sides and at least one side is Flagged by device.
  FN subject: A subject has one or two GT positive sides and none of these sides is Flagged by the device FP subject: A subject has both sides GT

CONTACTS AND LOCATIONS:
Locations (1):
- Solis Mammography Frisco at Stonebriar, Frisco, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided